CLINICAL TRIAL: NCT02603835
Title: A Multi-Center Evaluation of the Delivery of Intracoronary Hyperoxemic Supersaturated Oxygen Therapy for 60 Minutes in Anterior Acute Myocardial Infarction Patients With Successful Reperfusion (Via PCI) ≤ Six Hours After Symptom Onset
Brief Title: Evaluation of Intracoronary Hyperoxemic Oxygen Therapy in Anterior Acute Myocardial Infarction Patients (IC-HOT)
Acronym: IC-HOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TherOx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDE G120029/S007
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Anterior Wall Acute Myocardial Infarction
Keywords: SSO2 Therapy; Acute myocardial infarction; Anterior myocardial infarction; SuperSaturated oxygen delivery; Left main coronary artery; Myocardial infarction; Heart attack; Percutaneous coronary intervention; Cardiac catheterization laboratory; PCI; Stent; Stenting; Stents; Angioplasty; LMCA; Delivery of supersaturated oxygen (SSO2) therapy for the treatment of anterior acute myocardial infarction
MeSH Terms: conditions — Anterior Wall Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- SSO2 Therapy (Experimental): Delivery of SSO2 Therapy for 60 minutes selectively into the left main coronary artery (LMCA) using the TherOx DownStream System along with a single use disposable device called the TherOx DownStream Cartridge and a commercially available, qualified SSO2 delivery catheter
  Interventions: Device: SSO2 Therapy

INTERVENTIONS:
Device: SSO2 Therapy — Delivery of SSO2 Therapy for 60 minutes selectively into the left main coronary artery (LMCA) using the TherOx DownStream System along with a single use disposable device called the TherOx DownStream Cartridge and a commercially available, qualified SSO2 delivery catheter
  Other Names: TherOx DownStream System; TherOx DownStream Cartridge; SSO2 Delivery Catheter

SUMMARY:
The primary objective of the study is to collect confirmatory data supporting the safety and effectiveness of SSO2 Therapy in treatment of anterior acute myocardial infarction (AMI) patients who have undergone successful percutaneous coronary intervention (PCI) with stenting within six hours of experiencing AMI symptoms.

DETAILED DESCRIPTION:
A Multi-Center, Consecutively Enrolled Single-Arm Study to confirm the safety and effectiveness of the delivery of supersaturated oxygen (SSO2) Therapy for 60 minutes selectively into the left main coronary artery (LMCA) with a commercially available qualified SSO2 delivery catheter used with the TherOx® DownStream® System and Cartridge in the treatment of qualified patients presenting with anterior acute myocardial infarction in whom reperfusion with PCI is successful within six hours after symptom onset.

ELIGIBILITY:
GENERAL INCLUSION CRITERIA: Candidates for this study must meet ALL of the following criteria:

Pre-PCI:

1. The subject must be ≥18 and ≤80 years of age.
2. AMI must be anterior (ST-segment elevation >1 mm in two or more contiguous leads between V1 and V4 or new left bundle branch block).
3. Subject is experiencing clinical symptoms consistent with anterior AMI of ≤6 hour duration from time of symptom onset until admission to the emergency room.
4. The subject or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided and signed written informed consent, approved by the appropriate Institutional Review Board (IRB).
5. Subject and his/her physician agree to all required follow-up procedures and visits.

   ANGIOGRAPHIC INCLUSION CRITERIA: These are evaluated after the subject has provided signed informed consent but prior to enrollment:
6. Based on coronary anatomy, PCI is indicated for revascularization of the culprit lesion(s) with use of a commercially available coronary stent (bare metal or drug-eluting, at operator discretion) in the LAD.
7. The primary stented infarct-related lesion(s) must be in the proximal and/or mid-LAD coronary artery (other lesions in the LAD target vessel, including diagonal branches, may be treated if clinically indicated).
8. Baseline (pre-PCI) TIMI flow grade 0, 1, 2, or 3 flow in the LAD.
9. Successful angioplasty as documented by <50% diameter residual angiographic stenosis within all treated culprit lesions with TIMI 2 or 3 flow and no major complications such as perforation or shock.
10. Expected ability to place the SSO2 delivery catheter in the coronary ostium of the left main coronary system to deliver SSO2 Therapy with stable, coaxial alignment.

GENERAL EXCLUSION CRITERIA:

Pre-PCI:

1. Prior CABG surgery.
2. Prior myocardial infarction, or known prior systolic dysfunction (known ejection fraction <40% by any prior measure or regional wall motion abnormalities; this criterion does not include left ventricular dysfunction induced by the acute MI).
3. Thrombolytic therapy administered for this STEMI.
4. An elective surgical procedure is planned that would necessitate interruption of anti-platelet agents during the first 30 days post-enrollment.
5. Subjects who previously underwent coronary stent implantation and in whom coronary angiography demonstrates stent thrombosis to be the cause of the anterior AMI.
6. Subjects who have previously undergone an angioplasty or stenting procedure in the left anterior descending coronary artery.
7. Subjects with ventricular pseudoaneurysm, VSD, or severe mitral valve regurgitation (with or without papillary muscle rupture).
8. Any contraindication to MRI imaging. This will include any of the following exclusions:

   * Cardiac pacemaker or implantable defibrillator;
   * Non-MRI compatible aneurysm clip;
   * Neural Stimulator (i.e., TENS unit);
   * Any implanted or magnetically activated device (insulin pump);
   * Any type of non-MRI compatible ear implant;
   * Metal shavings in the orbits;
   * Any metallic foreign body, shrapnel, or bullet in a location which the physician feels would present a risk to the subject;
   * Any history indicating contraindication to MRI, including claustrophobia or allergy to gadolinium;
   * Inability to follow breath hold instructions or to maintain a breath hold for >15 seconds; and
   * Known hypersensitivity or contraindication to gadolinium contrast.
9. Known impaired renal function (creatinine clearance <30 ml/min/1.73 m2
10. Known platelet count <100,000 cells/mm by the MDRD formula) or on dialysis. 3 or >700,000 cells/mm3
11. Subject has active bleeding or a history of bleeding diathesis or coagulopathy (including heparin induced thrombocytopenia), or refusal to receive blood transfusions if necessary. or a known Hgb <10 g/dL.
12. History of intracerebral mass, aneurysm, arteriovenous malformation, or hemorrhagic stroke.
13. Stroke or transient ischemic attack within the past six (6) months, or any permanent neurological defect.
14. Gastrointestinal or genitourinary bleeding within the last two (2) months, or any major surgery (including CABG) within six weeks of enrollment.
15. Subject has received any organ transplant or is on a waiting list for any organ transplant.
16. Subject has other medical illness (e.g., cancer, dementia) or known history of substance abuse (alcohol, cocaine, heroin, etc.) that may cause non-compliance with the protocol, confound the data interpretation, or is associated with limited life expectancy of less than one year.
17. Subject has a known hypersensitivity or contraindication to unfractionated heparin, abciximab, aspirin, bivalirudin, cangrelor, clopidogrel, ticlopidine, prasugrel, or ticagrelor that cannot be adequately premeditated.
18. Current use of warfarin, dabigatran, or factor Xa inhibitors, or known intent to administer these agents after the primary PCI.
19. Subjects presenting with or developing in the cath lab prior to completion of the primary PCI procedure any of the following conditions: cardiogenic shock (SBP <80 mmHg for >30 minutes), or requiring IV pressors or emergent placement of an intra-aortic balloon pump (IABP), Impella, or other hemodynamic support for hypotension treatment, or cardiopulmonary resuscitation for >10 minutes, or ventricular fibrillation or tachycardia requiring cardioversion or defibrillation.
20. Severe known cardiac valvular stenosis or insufficiency, pericardial disease, or non-ischemic cardiomyopathy.
21. Any significant medical or social condition which in the investigator's opinion may interfere with the subject's participation in the study or ability to comply with follow-up procedures, including MRI (e.g. alcoholism, dementia, lives far from the research center, etc.).
22. Current participation in other investigational device or drug trials that have not finished the primary endpoint follow-up period.
23. Previous enrollment in this study.

    ANGIOGRAPHIC EXCLUSION CRITERIA: These are evaluated after the subject has provided signed Informed Consent but prior to enrollment:
24. Anticipated inability to achieve a stable coaxial position in the left main coronary artery with the SSO2 delivery catheter.
25. Treatment during the index procedure of any lesion in either the left main, LCX (including the ramus), and/or RCA.
26. Post-index procedure planned intervention within 30 days (i.e., PCI of non-target lesions in any vessel, or CABG). Note: Planned revascularization (PCI or bypass) of a non-target lesion >30 days following the index procedure is allowed.
27. Anterior MI is due to thrombosis within or adjacent to a previously implanted stent.
28. Left ventriculography demonstrates severe mitral regurgitation, a ventricular septal defect, or a pseudoaneurysm.
29. Any left main coronary artery stenosis >20%.
30. Any untreated LAD or diagonal branch lesion is present with diameter stenosis > 50% in a vessel with reference vessel diameter > 2.0 mm (visually estimated), or for which PCI will be required before the MRI study.
31. Presence of a non-stented coronary dissection with NHLBI grade >B upon completion of the PCI procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W. Stone, MD, Principal Investigator — Columbia University
Locations (15):
- United States (15):
  - Heart Center, Inc., Huntsville, Alabama
  - Scripps Hospital, La Jolla, California
  - Danbury Hospital, Danbury, Connecticut
  - Alexian Brothers Heart & Vascular Institute, Elk Grove Village, Illinois
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Medical Center, Detroit, Michigan
  - St. John Hospital & Medical Center, Detroit, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Providence-Providence Park Hospital, Southfield, Michigan
  - WakeMed Heart Center, Raleigh, North Carolina
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Holy Spirit Cardiology, Camp Hill, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - The Miriam Hospital/Rhode Island Hospital, Providence, Rhode Island
  - Wellmont CVA Heart Institute, Kingsport, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen S, David SW, Khan ZA, Metzger DC, Wasserman HS, Lotfi AS, Hanson ID, Dixon SR, LaLonde TA, Genereux P, Ozan MO, Maehara A, Stone GW. One-year outcomes of supersaturated oxygen therapy in acute anterior myocardial infarction: The IC-HOT study. Catheter Cardiovasc Interv. 2021 May 1;97(6):1120-1126. doi: 10.1002/ccd.29090. Epub 2020 Jul 10. PMID 32649037

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SSO2 Therapy
Started | 100
Completed | 93
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | SSO2 Therapy
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 96
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 91
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Net Adverse Clinical Events (NACE)
Description: Composite of death, reinfarction, clinically-driven target vessel revascularization, stent thrombosis (ARC definite or probable), new onset severe heart failure or readmission for heart failure, and TIMI major or minor bleeding. This outcome measure includes a hierarchical sum of the events, meaning if a subject experiences two event types they are only counted once in the overall NACE rate.
Time Frame: 30-Day
Population: All treated subjects
Measure: Count of Participants; unit: Participants
Arm/Group | SSO2 Therapy
Number analyzed (Participants) | 98
Participants
  Overall NACE | 7
  Death | 0
  Reinfarction/Spontaneous MI | 1
  Clinically Driven Target Vessel Revascularization | 1
  TIMI Major or Minor Bleeding | 4
  New Onset Severe Heart Failure | 1
  ARC Definite/Probable Stent Thrombosis | 1

2. Secondary Outcome: Rate of Target Lesion Failure
Description: Composite of cardiac death , target vessel MI, or clinically driven target Lesion revascularization
Time Frame: 30 days
Population: All treated subjects
Measure: Count of Participants; unit: Participants
Arm/Group | SSO2 Therapy
Number analyzed (Participants) | 98
Participants | 1

3. Secondary Outcome: Rate of Net Adverse Clinical Events (NACE)
Description: Composite of death, reinfarction, clinically-driven target vessel revascularization, stent thrombosis (ARC definite or probable), new onset severe heart failure or readmission for heart failure, and TIMI major or minor bleeding. This outcome measure includes a hierarchical sum of the events, meaning if a subject experiences two or more event types they are only counted once in the overall NACE rate.
Time Frame: 1 year
Population: All treated subjects population (n=100) minus subjects that discontinued the study prior to the 12-month follow-up (n=7).
Measure: Count of Participants; unit: Participants
Arm/Group | SSO2 Therapy
Number analyzed (Participants) | 93
Participants
  Overall NACE | 10
  Death | 0
  Reinfarction/Spontaneous MI | 3
  Clinically Driven Target Vessel Revascularization | 3
  TIMI Major or Minor Bleeding | 5
  New Onset Severe Heart Failure | 1
  ARC Definite/Probable Stent Thrombosis | 1

4. Secondary Outcome: Target Lesion Failure
Description: Composite of cardiac death , target vessel MI, or clinically driven target Lesion revascularization
Time Frame: 1 year
Population: All Treated Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | SSO2 Therapy
Number analyzed (Participants) | 100
Participants | 3

5. Secondary Outcome: Median Infarct Size by Cardiac MRI
Description: Measurement of the % left ventricle (LV) necrosis
Time Frame: 30 days
Population: All treated subjects with analyzable cardiac MRI scans
Measure: Median (Inter-Quartile Range); unit: percentage of myocardial mass
Arm/Group | SSO2 Therapy
Number analyzed (Participants) | 85
percentage of myocardial mass | 19.4 [8.8 to 28.9]

6. Secondary Outcome: Microvascular Obstruction by Cardiac MRI
Description: Measurement of the % left ventricle (LV) showing microvascular obstruction
Time Frame: 4 days post-procedure
Population: All treated subjects with analyzable cardiac MRI scans
Measure: Median (Inter-Quartile Range); unit: percentage of MVO of myocardial mass
Arm/Group | SSO2 Therapy
Number analyzed (Participants) | 78
percentage of MVO of myocardial mass | 0.30 [0.0 to 2.4]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were reported throughout the trial for all subjects, including at each protocol-specified follow-up assessment period, i.e., post-index procedure, hospital discharge, 30-day follow-up, 6-month follow-up and 1 year follow-up.
Arm/Group | SSO2 Therapy
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 27/100
Other Adverse Events (participants affected / at risk) | 68/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSO2 Therapy (N=100)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2)
Angina Pectoris (Cardiac disorders) | 4 (4)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1)
Torsade de Pointes (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Vascular Injury (Injury, poisoning and procedural complications) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Percutaneous Coronary Intervention (Surgical and medical procedures) | 1 (1)
Aortic Valve Replacement (Surgical and medical procedures) | 1 (1)
Coronary Artery Bypass (Surgical and medical procedures) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Aortic Stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSO2 Therapy (N=100)
Angina Pectoris (Cardiac disorders) | 17 (18)
Cardiac Failure Congestive (Cardiac disorders) | 9 (9)
Atrial Fibrillation (Cardiac disorders) | 5 (5)
Fatigue (General disorders) | 6 (6)
Dizziness (Cardiac disorders) | 4 (4)
Ventricular Tachycardia (Cardiac disorders) | 4 (4)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3)
Cardiac Ventricular Thrombosis (Cardiac disorders) | 3 (3)
Ischaemic Cardiomyopathy (Cardiac disorders) | 3 (3)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Dyspnoea (Cardiac disorders) | 2 (2)
Dyspnoea Exertional (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Syncope (Cardiac disorders) | 2 (2)
Arteriospasm Coronary (Cardiac disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Presyncope (Cardiac disorders) | 1 (1)
Pulmonary Oedema (Cardiac disorders) | 1 (1)
Sinus Arrest (Cardiac disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Torsade de Pointes (Cardiac disorders) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Ventricular Hypokinesia (Cardiac disorders) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Vision Blurred (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Consitpation (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 3 (3)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vascular Stent Thrombosis (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Acute Sinusitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection Fungal (Infections and infestations) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Periorbital Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular Injury (Injury, poisoning and procedural complications) | 1 (1)
Blood Electrolytes Abnormal (Investigations) | 1 (1)
Ejection Fraction Decreased (Investigations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Device Operational Issue (Product Issues) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic Valve Replacement (Surgical and medical procedures) | 1 (1)
Coronary Artery Bypass (Surgical and medical procedures) | 1 (1)
Mitral Valve Replacement (Surgical and medical procedures) | 1 (1)
Percutaneous Coronary Intervention (Surgical and medical procedures) | 1 (1)
Haematoma (Vascular disorders) | 6 (6)
Hypotension (Vascular disorders) | 6 (6)
Haemorrhage (Vascular disorders) | 5 (6)
Hypertension (Vascular disorders) | 2 (2)
Aortic Stenosis (Vascular disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the clinical trial agreement executed between the Sponsor and one or more Primary Investigators:

"The PRIMARY INVESTIGATOR and/or other INSTITUTION clinical research personnel cannot publicly report the single-center results until an all-inclusive multicenter manuscript is in press or one (1) year following the completion of this STUDY."

DOCUMENTS (2):
  • Study Protocol (2015-11-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT02603835/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT02603835/SAP_001.pdf